CLINICAL TRIAL: NCT04376411
Title: Possible Role of Regulatory B Cells in Behçet's Disease: Special Interest in Cardiovascular System
Brief Title: Role of Regulatory B Cells in Behçet's Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, safaa Mahran, Associate Proffesor, Assiut University
Other Study IDs: 17300388
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Behcet Disease
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with Behcet disease: Flow-cytometric assay Detailed 2 Di mention Echocardiographic analysis Two-Dimensional speckle tracking echocardiography
  Interventions: Diagnostic Test: Flow-cytometric assay; Diagnostic Test: 2D Echocardiographic analysis; Diagnostic Test: Two-Dimensional speckle tracking echocardiography
- Healthy control subjects: Flow-cytometric assay
  Interventions: Diagnostic Test: Flow-cytometric assay

INTERVENTIONS:
Diagnostic Test: Flow-cytometric assay — 100 µl of blood sample was incubated for 20 minutes at 4 C in the dark. Following incubation, red blood cells lysis, washing and analysis a specific software.Forward and side scatter histogram was used to define the lymphocytes population.
Diagnostic Test: 2D Echocardiographic analysis — Trans thoracic echocardiographic examination was performed through (PHILIPS -33) echocardiography device with broadband S5-1 transducer
  Groups: patients with Behcet disease
Diagnostic Test: Two-Dimensional speckle tracking echocardiography — Two-Dimensional speckle tracking echocardiography was performed on grey scale images of the left ventricle. For offline analysis digital storage software (Qlab 10.4) was used. The frame rate was adjusted to be 60-90 frame/second.
  Groups: patients with Behcet disease

SUMMARY:
There are limited data about the role of regulatory B cells in Behcet Disease. In this study we aimed to identify the proportions of total B lymphocytes and their regulatory subset in different Behcet Disease phenotype and therapies concentrating on the cardiovascular system attempting to unravel their function in Behcet Disease.

DETAILED DESCRIPTION:
Behçet's disease is a chronic multi-organ vasculitis characterized by recurrent oral and genital aphthae, skin lesions, widespread thrombosis and aneurysmal formation, and serious involvement of the eyes and central nervous system.

The innate and adaptive immune cells integrate in the pathogenesis of Behçet's disease. Interestingly, the gene expression analysis of Behçet's disease patients and healthy controls revealed the modulation of a range of genes involved in biological processes in Behçet's disease such as inflammation, apoptosis, angiogenesis, blood coagulation, vascular damage, signalling pathways, and immune responses, particularly, in innate immune cells, Th17 cells and B cells. Yet, the regulatory role of B cells in Behçet's disease has not been thoroughly investigated. Therefore, the aim of the current study is to identify the proportions of total B lymphocytes and their regulatory subset in different Behçet's disease phenotypes and therapies attempting to unravel their function in Behcet Disease. The role of B cells and regulatory B cells in the cardiovascular system affection in Behcet Disease was studied in more details.

ELIGIBILITY:
Inclusion Criteria:

* Thirty five adult patients who fulfilled the diagnostic criteria of Behcet Disease, and 39 age and sex matched healthy subjects as control

Exclusion Criteria:

* Patients younger than 18 years old and those who were affected by other rheumatic disease other than Behcet Disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty five adult patients who fulfilled the diagnostic criteria of Behcet Disease, and 39 age and sex matched healthy subjects as control
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
percentage of B and B regulatory cells in different Behcet phenotype | 1 day (done once)
  correlation between the B and B regulatory cells with different presentations of Behcet disease especially the cardiovascular manifestations.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1- Kural-Seyahi E, Fresko I, Seyahi N, Ozyazgan Y, Mat C, Hamuryudan V, et al. The long-term mortality and morbidity of Behcet syndrome: a 2-decade outcome survey of 387 patients followed at a dedicated center. Medicine (Baltimore). 2003;82(1):60-76. 2- Kirino Y, Bertsias G, Ishigatsubo Y, Mizuki N, Tugal-Tutkun I, Seyahi E, et al. Genome-wide association analysis identifies new susceptibility loci for Behcet's disease and epistasis between HLA-B*51 and ERAP1. Nat Genet. 2013;45(2):202-7. 3- Yoon JY, Lee Y, Yu SL, Yoon HK, Park HY, Joung CI, et al. Aberrant expression of interleukin-10 and activation-induced cytidine deaminase in B cells from patients with Behcet's disease. Biomed Rep. 2017;7(6):520-6.